CLINICAL TRIAL: NCT00265122
Title: A Multicenter, Randomized, Phase 2a Study of Human Monoclonal Antibody to IL-12p40 (CNTO 1275) in Subjects With Moderately to Severely Active Crohn's Disease
Brief Title: A Study of the Safety and Efficacy of Ustekinumab (CNTO 1275) in Participants With Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR005287; C0379T07 (Other: Centocor, Inc.)
Record Dates: First submitted 2005-12-13; First posted 2005-12-14 (Estimated); Results first posted 2013-07-31 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-01

CONDITIONS: Crohn Disease
Keywords: Crohn Disease; Biologic; Infusion; Injection; CNTO 1275; Ustekinumab; C01275; IL-12p40
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Population 1: Placebo SC followed by ustekinumab SC (Experimental): Placebo injected subcutaneously (SC) once a week for 4 weeks (Weeks 0-3) during Intervention Period 1 followed by ustekinumab 90 mg SC once a week for 4 weeks (Weeks 8-11) during Intervention Period 2.
  Interventions: Drug: Ustekinumab 90 mg; Drug: Placebo SC
- Population 1: Ustekinumab SC followed by Placebo SC: (Experimental): Ustekinumab 90 mg injected subcutaneously (SC) once a week for 4 weeks (Weeks 0-3) during Intervention Period 1 followed by ustekinumab 90 mg SC once a week for 4 weeks (Weeks 8-11) during Intervention Period 2.
  Interventions: Drug: Ustekinumab 90 mg; Drug: Placebo SC
- Population 1: Placebo IV followed by ustekinumab IV (Experimental): Placebo given as 1 intravenous (IV) infusion at Week 0 during Intervention Period 1 and ustekinumab 4.5 mg/kg given as one IV infusion at Week 8 during Intervention Period 2.
  Interventions: Drug: Ustekinumab 4.5 mg/kg; Drug: Placebo IV
- Population 1: Ustekinumab IV followed by Placebo IV: (Experimental): Ustekinumab 4.5 mg/kg given as one intravenous(IV) infusion at Week 0 during Intervention Period 1 followed by placebo given as one IV infusion at Week 8 during Intervention Period 2.
  Interventions: Drug: Ustekinumab 4.5 mg/kg; Drug: Placebo IV
- Population 2: Ustekinumab SC (Experimental): Ustekinumab 90 mg injected subcutaneously (SC) once a week at Weeks 0-3 during Intervention Period 1. No intervention given during Intervention Period 2.
  Interventions: Drug: Ustekinumab 90 mg
- Population 2: Ustekinumab IV (Experimental): Ustekinumab 4.5 mg given as one intravenous (IV) infusion at Week 0 during Intervention Period 1. No intervention given during Intervention Period 2.
  Interventions: Drug: Ustekinumab 4.5 mg/kg

INTERVENTIONS:
Drug: Ustekinumab 90 mg — one 90 mg SC injection each week for 4 weeks (Weeks 0-3 during Intervention Period 1 or Weeks 8-11 during Intervention Period 2 for Population 1 or Weeks 0-3 during Intervention Period 1 for Population 2)
  Other Names: CNTO 1275
  Arms: Population 1: Placebo SC followed by ustekinumab SC; Population 1: Ustekinumab SC followed by Placebo SC:; Population 2: Ustekinumab SC
Drug: Ustekinumab 4.5 mg/kg — one IV infusion of 4.5 mg/kg over a period of not less than 2 hours at Week 0 in Intervention Period 1 or Week 8 in Intervention Period 2 for Population 1 or at Week 0 in Intervention Period 1 for Population 2
  Other Names: CNTO 1275
  Arms: Population 1: Placebo IV followed by ustekinumab IV; Population 1: Ustekinumab IV followed by Placebo IV:; Population 2: Ustekinumab IV
Drug: Placebo SC — one SC injection each week for 4 weeks (Weeks 0-3 in Intervention Period 1 or Weeks 8-11 in Intervention Period 2 for Population 1 or at Weeks 0-3 in Intervention Period 1 for Population 2)
  Arms: Population 1: Placebo SC followed by ustekinumab SC; Population 1: Ustekinumab SC followed by Placebo SC:
Drug: Placebo IV — one IV infusion over a period of not less than 2 hours at Week 0 in Intervention Period 1 for Population 1 and Population 2 or at Week 8 in Intervention Period 2 for Population 1
  Arms: Population 1: Placebo IV followed by ustekinumab IV; Population 1: Ustekinumab IV followed by Placebo IV:

SUMMARY:
The purpose of this study is to examine the safety and efficacy of CNTO 1275 in participants with active Crohn's Disease.

DETAILED DESCRIPTION:
This is a multicenter, randomized study of IL-12p40 (CNTO 1275), hereafter referred to as ustekinumab, in 2 populations of participants with moderately to severely active Crohn's disease of at least 6 weeks duration. A total of approximately 120 volunteers will participate in this study in Canada, Belgium, and the United States. Two separate groups of participants (Population 1 and Population 2) will be evaluated. The primary population of participants (Population 1) will consist of approximately 100 participants with Crohn's disease despite treatment with standard Crohn's disease medications (includes agents to decrease intestinal inflammation such as 5-ASA medications such as PENTASA, ASACOL), corticosteroids such as prednisone and/or other drugs known to suppress the immune system called immunomodulators such as azathioprine, 6-mercaptopurine, methotrexate, infliximab or adalimumab [marketed under the trade name of HUMMIRA]). Participants in Population 1 will be randomly assigned (assigned by chance, like "flipping a coin") to double-blind treatment (participants and study staff will not know the identity of the treatments) with ustekinumab and placebo (inactive substance) in 1 of 4 treatment groups as follows: (1) 4 weeks of treatment with ustekinumab 90 mg followed by 4 weeks of treatment with placebo injected subcutaneously (SC, under the skin), (II) 4 weeks of placebo followed by 4 weeks of ustekinumab 90 mg injected SC, (III) 1 intravenous (IV, in the vein) infusion of ustekinumab 4.5 mg/kg followed by 1 IV infusion of placebo, and (IV) 1 IV infusion of placebo followed by 1 IV infusion of ustekinumab 4.5 mg/kg. Population 2 consists of approximately 20 participants who failed to respond to previous therapy with infliximab (trade name REMICADE), a type of antibody that decreases inflammation in patients with moderate to severe Crohn's disease). All participants in Population 2 will receive open-label (un-blinded) treatment with ustekinumab 4.5 mg/kg administered SC for 4 weeks or as one IV infusion. Placebo will not be given to participants in Population 2. The duration of the study for each participant is 28 weeks (not including a screening period of up to 2 weeks) with participants returning at Week 54 to have blood samples collected to assess the concentration of ustekinumab and antibodies to ustekinumab. Adverse events (side-effects) as a measure of safety and tolerability and results from routine laboratory tests will be monitored and reported throughout the study from the time that informed consent is documented up to 3 days after the final blood sample collection at Week 54. Note: doses of ustekinumab used in the study were adjusted by a factor of 0.9 to be consistent with the corrected absorptivity constant for ustekinumab. Therefore, ustekinumab doses of 100 mg and 5 mg/kg previously stated in the study protocol have been restated as 90 mg and 4.5 mg/kg, respectively. No change was made to the amount of ustekinumab given to participants in this study.

ELIGIBILITY:
Inclusion Criteria:

* Have moderately to severly active Crohn's disease or fistulizing Crohn's disease for at least 6 weeks' duration with a Crohn's disease activity index (CDAI) score of >=220 and <=450
* In Population 1, participants must have had active disease despite treatment with 5-ASA compounds, antibiotics, corticosteroids, and/or immunomodulators, including anti-TNF agents. In Population 2, participants must have had active disease and have failed to respond to infliximab at the maximum approved dose and treatment regimen for Crohn's disease as defined in the US package insert.

Exclusion Criteria:

* Have local manifestations of Crohn's disease such as strictures, abscesses, or other disease complications for which surgery might be indicated
* Had intra-abdominal surgery within 6 months prior to entering the study
* Have received treatment with parenteral nutrition (ie, introduction of nutrition into the body via a route other than the mouth) (total parenteral nutrition [TPN]) within 6 weeks of baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2004-04; Primary Completion 2005-11 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor Clinical Trial, Study Director — Centocor, Inc.
Locations (57):
- United States (50):
  - Scottsdale, Arizona
  - Anaheim, California
  - Sacramento, California
  - San Francisco, California
  - Bristol, Connecticut
  - New Haven, Connecticut
  - Jacksonville, Florida
  - Miami, Florida
  - Indianapolis, Indiana
  - Topeka, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Metairie, Louisiana
  - New Orleans, Louisiana
  - Laurel, Maryland
  - Chesterfield, Michigan
  - Troy, Michigan
  - Rochester, Minnesota
  - Omaha, Nebraska
  - Great Neck, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Beaver Falls, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Columbia, South Carolina
  - Germantown, Tennessee
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Ogden, Utah
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Christiansburg, Virginia
  - Richmond, Virginia
  - Everett, Washington
  - Seattle, Washington
  - Tacoma, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Leuven, Belgium
- Canada (6):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Toronto, Ontario
  - Hamilton
  - London

REFERENCES:
- [Derived] Ghosh S, Gensler LS, Yang Z, Gasink C, Chakravarty SD, Farahi K, Ramachandran P, Ott E, Strober BE. Ustekinumab Safety in Psoriasis, Psoriatic Arthritis, and Crohn's Disease: An Integrated Analysis of Phase II/III Clinical Development Programs. Drug Saf. 2019 Jun;42(6):751-768. doi: 10.1007/s40264-019-00797-3. PMID 30739254
- [Derived] Sandborn WJ, Feagan BG, Fedorak RN, Scherl E, Fleisher MR, Katz S, Johanns J, Blank M, Rutgeerts P; Ustekinumab Crohn's Disease Study Group. A randomized trial of Ustekinumab, a human interleukin-12/23 monoclonal antibody, in patients with moderate-to-severe Crohn's disease. Gastroenterology. 2008 Oct;135(4):1130-41. doi: 10.1053/j.gastro.2008.07.014. Epub 2008 Jul 17. PMID 18706417

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 131 participants (104 in Population 1 and 27 in Population 2) were enrolled among 42 study centers (35 centers in the US, 6 in Canada, and 1 in Belgium) to receive treatment with placebo or ustekinumab (CNTO 1275) administered subcutaeously (injected under the skin [SC]) or intravenously (infused in a vein [IV]).
Pre-assignment Details: Participants with moderate to severe active Crohn's Disease despite treatment with 5-ASA compounds, antibiotics, corticosteroids, and/or immunomodulators, including anti-TNF agents were enrolled and referred to as Population 1 and those with active disease who failed to respond to infliximab were enrolled and referred to as Population 2.
Groups:
- Population 1: Ustekinumab 90 mg SC Followed by Placebo SC: Ustekinumab 90 mg injected subcutaneously (SC) once a week for 4 weeks (Weeks 0-3) during Intervention Period 1 followed by placebo SC once a week for 4 weeks (Weeks 8-11) during Intervention Period 2.
- Population 1: Placebo IV Followed by Ustekinumab 4.5 mg/kg IV: Placebo given as 1 intravenous (IV) infusion at Week 0 during Intervention Period 1 and ustekinumab 4.5 mg/kg given as one IV infusion at Week 8 during Intervention Period 2.
- Population 1: Ustekinumab 4.5 mg/kg IV Followed by Placebo IV: Ustekinumab 4.5 mg/kg given as one intravenous(IV) infusion at Week 0 during Intervention Period 1 followed by placebo given as one IV infusion at Week 8 during Intervention Period 2.
- Population 2: Ustekinumab 90 mg SC: Ustekinumab 90 mg injected subcutaneously (SC) once a week at Weeks 0-3 during Intervention Period 1. No intervention given during Intervention Period 2.
- Population 2: Ustekinumab 4.5 mg/kg IV: Ustekinumab 4.5 mg given as one intravenous (IV) infusion at Week 0 during Intervention Period 1. No intervention given during Intervention Period 2.
Period: Intervention Period 1 (Weeks 0 to 8):
Arm/Group | Population 1: Placebo SC Followed by Ustekinumab SC | Population 1: Ustekinumab 90 mg SC Followed by Placebo SC | Population 1: Placebo IV Followed by Ustekinumab 4.5 mg/kg IV | Population 1: Ustekinumab 4.5 mg/kg IV Followed by Placebo IV | Population 2: Ustekinumab 90 mg SC | Population 2: Ustekinumab 4.5 mg/kg IV
Started | 26 | 25 | 27 | 26 | 14 | 13
Completed | 24 | 23 | 22 | 24 | 13 | 13
Not Completed | 2 | 2 | 5 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 3 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 1 | 2 | 1 | 0 | 0
Period: Intervention Period 2 (Weeks 8 to 28):
Arm/Group | Population 1: Placebo SC Followed by Ustekinumab SC | Population 1: Ustekinumab 90 mg SC Followed by Placebo SC | Population 1: Placebo IV Followed by Ustekinumab 4.5 mg/kg IV | Population 1: Ustekinumab 4.5 mg/kg IV Followed by Placebo IV | Population 2: Ustekinumab 90 mg SC | Population 2: Ustekinumab 4.5 mg/kg IV
Started | 24 | 23 | 22 | 24 | 13 | 13
Completed | 17 | 22 | 18 | 20 | 8 | 12
Not Completed | 7 | 1 | 4 | 4 | 5 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 3 | 1 | 3 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 2 | 2 | 1
Not completed — Other | 4 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Population 1: Placebo SC Followed by Ustekinumab SC | Population 1: Ustekinumab 90 mg SC Followed by Placebo SC | Population 1: Placebo IV Followed by Ustekinumab 4.5 mg/kg IV | Population 1: Ustekinumab 4.5 mg/kg IV Followed by Placebo IV | Population 2: Ustekinumab 90 mg SC | Population 2: Ustekinumab 4.5 mg/kg IV | Total
Number analyzed (Participants) | 26 | 25 | 27 | 26 | 14 | 13 | 131
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.7 (13.99) | 36.5 (13.17) | 43.5 (11.39) | 43.1 (12.23) | 46.9 (13.63) | 42.7 (11.27) | 40.0 (12.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 14 | 12 | 6 | 8 | 61
  Male | 15 | 15 | 13 | 14 | 8 | 5 | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Population 1 With a Clinical Response at Week 8
Description: The table below provides the number of participants in Population 1 with a clinical response at Week 8 defined as a reduction from baseline in the CDAI (Crohn's disease activity index) score of >= 25% and >= 70 points at Week 8. A reduction in CDAI score correlates with improvement in the severity of illness. The CDAI is derived as a weighted sum of 8 different Crohn's disease related variables: extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools (or bags emptied for participants with a stoma), abdominal pain/cramping, use of antidiarrheal drug(s) and/or opiates, and general well being. The primary endpoint analysis was based on the comparison between the combined SC and IV Placebo and combined SC and IV ustekinumab treatment groups in Population 1.
Time Frame: Week 8
Population: The analysis included all randomized patients (ITT), regardless of whether they had any protocol deviations.
Measure: Number; unit: participants
Groups:
- Population 1: Placebo SC and IV Combined: All particpants who received Placebo SC and Placebo IV
- Population 1: Ustekinumab SC and IV Combined: All participants who received Ustekinumab 90 mg SC and Ustekinumab 4.5 mg/kg IV
Arm/Group | Population 1: Placebo SC Followed by Ustekinumab SC | Population 1: Ustekinumab 90 mg SC Followed by Placebo SC | Population 1: Placebo IV Followed by Ustekinumab 4.5 mg/kg IV | Population 1: Ustekinumab 4.5 mg/kg IV Followed by Placebo IV | Population 1: Placebo SC and IV Combined | Population 1: Ustekinumab SC and IV Combined
Number analyzed (Participants) | 26 | 25 | 27 | 26 | 53 | 51
participants | 13 | 12 | 8 | 13 | 21 | 25
Statistical Analysis 1: Comparison: Population 1: Placebo SC and IV Combined vs Population 1: Ustekinumab SC and IV Combined; Null hypothesis: No difference between ustekinumab and placebo at a significant level of 0.05; Test type: Superiority or Other; p = 0.337, Cochran-Mantel-Haenszel — The P-Value is from a Cochran-Mantel-Haenszel (CMH) test stratified by the route of administration

2. Secondary Outcome: Number of Participants in Population 2 With a Clinical Response at Week 8
Description: The table below provides the number of participants in Population 2 with a clinical response at Week 8 defined as a reduction from baseline in the CDAI (Crohn's disease activity index) score of >= 25% and >= 70 points at Week 8. A reduction in CDAI score correlates with improvement in the severity of illness. The CDAI is derived as a weighted sum of 8 different Crohn's disease related variables: extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools (or bags emptied for participants with a stoma), abdominal pain/cramping, use of antidiarrheal drug(s) and/or opiates, and general well-being.
Time Frame: Week 8
Population: The analysis included all randomized patients (ITT), regardless of whether they had any protocol deviations.
Measure: Number; unit: participants
Groups:
- Population 2: Ustekinumab 90 SC: Paticipants received ustekinumab 90 mg subcutaneously (SC) at Weeks 0, 1, 2, and 3 (Intervention Period 1: Weeks 0-8), and did not receive any study agent from Week 8 onward (Intervention Period 2: Weeks 8-28)
Arm/Group | Population 2: Ustekinumab 90 SC | Population 2: Ustekinumab 4.5 mg/kg IV
Number analyzed (Participants) | 14 | 13
participants | 6 | 7

3. Secondary Outcome: Number of Participants in Population 1 With Clinical Remission at Week 8
Description: The table below shows the number of participants in Population 1 with clinical remission at Week 8 defined a CDAI (Crohn's disease activity index) score < 150 points at Week 8. A reduction in CDAI score correlates with improvement in the severity of illness. The CDAI is derived as a weighted sum of 8 different Crohn's disease related variables: extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools (or bags emptied for participants with a stoma), abdominal pain/cramping, use of antidiarrheal drug(s) and/or opiates, and general well-being.
Time Frame: Week 8
Population: The analysis included all randomized patients (ITT), regardless of whether they had any protocol deviations.
Measure: Number; unit: participants
Groups:
- Population 1:Placebo SC Followed by Ustekinumab 90 mg SC: Participants received subcutaneous (SC) injections of placebo at Weeks 0, 1, 2, 3 (Intervention Period 1: Weeks 0-8), and 90 mg ustekinumab SC at Weeks 8, 9, 10 and 11 (Intervention Period 2: Weeks 8-28)
- Population 1: Placebo SC and IV Combined: All participants who received Placebo SC and Placebo IV
- Population 1: Ustekinumab SC and IV Combined: All participants who received Ustekinumab SC and Ustekinumab IV
Arm/Group | Population 1:Placebo SC Followed by Ustekinumab 90 mg SC | Population 1: Ustekinumab 90 mg SC Followed by Placebo SC | Population 1: Placebo IV Followed by Ustekinumab 4.5 mg/kg IV | Population 1: Ustekinumab 4.5 mg/kg IV Followed by Placebo IV | Population 1: Placebo SC and IV Combined | Population 1: Ustekinumab SC and IV Combined
Number analyzed (Participants) | 26 | 25 | 27 | 26 | 53 | 51
participants | 6 | 6 | 3 | 7 | 9 | 13
Statistical Analysis 1: Comparison: Population 1: Placebo SC and IV Combined vs Population 1: Ustekinumab SC and IV Combined; Test type: Superiority or Other; p = 0.292, Cochran-Mantel-Haenszel — The P-Value is from a CMH test stratified by the route of administration

ADVERSE EVENTS:
Time Frame: Week 28
Description: The number of participants at risk for adverse events was based on actual treatment received which differs from the number of participants randomized to treatment reported in Participant flow. Adverse events following the first administration of ustekinumab are included in the table.
Groups:
- Population 1: Placebo SC Followed by Ustekinumab SC: Placebo injected subcutaneously (SC) once a week for 4 weeks (Weeks 0-3) during Intervention Period 1 followed by ustekinumab 90 mg SC once a week for 4 weeks (Weeks 8-11) during Intervention Period 2. NOTE: 4 of 26 participants randomized to this treatment group received placebo only and were excluded from the "Total # at Risk by any Serious Adverse Event" and "Total # at Risk by any Other Adverse Event" listed below.
- Population 1: Placebo IV Followed by Ustekinumab 4.5 mg/kg IV: Placebo given as 1 intravenous (IV) infusion at Week 0 during Intervention Period 1 and ustekinumab 4.5 mg/kg given as one IV infusion at Week 8 during Intervention Period 2. NOTE: 8 of 27 participants randomized to this treatment group were excluded from the "Total # at Risk by any Serious Adverse Event" and "Total # at Risk by any Other Adverse Event" listed below for the following reasons: 7 participants received placebo only were excluded from the analysis of adverse events and 1 participant received ustekinumab IV at Week 0 and was included in the analysis of adverse events in the treatment group labelled "Ustekinumab 4.5 mg/kg IV followed by Placebo IV."
- Population 1: Ustekinumab 4.5 mg/kg IV Followed by Placebo IV: Ustekinumab 4.5 mg/kg given as one intravenous(IV) infusion at Week 0 during Intervention Period 1 followed by placebo given as one IV infusion at Week 8 during Intervention Period 2. NOTE: 26 participants randomized to this treatment group + 1 participant randomized to treatment with "Placebo IV followed by Ustekinumab 4.5 mg/kg IV" who received ustekinumab IV at Week 0 was included in the "Total # at Risk by any Serious Adverse Event" and "Total # at Risk by any Other Adverse Event" listed below.
Arm/Group | Population 1: Placebo SC Followed by Ustekinumab SC | Population 1: Ustekinumab 90 mg SC Followed by Placebo SC | Population 1: Placebo IV Followed by Ustekinumab 4.5 mg/kg IV | Population 1: Ustekinumab 4.5 mg/kg IV Followed by Placebo IV | Population 2: Ustekinumab 90 mg SC | Population 2: Ustekinumab 4.5 mg/kg IV
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/25 | 2/19 | 3/27 | 2/14 | 2/13
Other Adverse Events (participants affected / at risk) | 16/22 | 23/25 | 16/19 | 21/27 | 12/14 | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Population 1: Placebo SC Followed by Ustekinumab SC (N=22) | Population 1: Ustekinumab 90 mg SC Followed by Placebo SC (N=25) | Population 1: Placebo IV Followed by Ustekinumab 4.5 mg/kg IV (N=19) | Population 1: Ustekinumab 4.5 mg/kg IV Followed by Placebo IV (N=27) | Population 2: Ustekinumab 90 mg SC (N=14) | Population 2: Ustekinumab 4.5 mg/kg IV (N=13)
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Histoplasmosis disseminated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Colonic stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Population 1: Placebo SC Followed by Ustekinumab SC (N=22) | Population 1: Ustekinumab 90 mg SC Followed by Placebo SC (N=25) | Population 1: Placebo IV Followed by Ustekinumab 4.5 mg/kg IV (N=19) | Population 1: Ustekinumab 4.5 mg/kg IV Followed by Placebo IV (N=27) | Population 2: Ustekinumab 90 mg SC (N=14) | Population 2: Ustekinumab 4.5 mg/kg IV (N=13)
Nausea (Gastrointestinal disorders) | 5 | 2 | 2 | 3 | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 0 | 5 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 0 | 3 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 0 | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bowel sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intestinal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Spigelian hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 6 | 4 | 4 | 7 | 4 | 4
Upper respiratory tract infection (Infections and infestations) | 6 | 5 | 3 | 4 | 1 | 3
Nasopharyngitis (Infections and infestations) | 1 | 3 | 1 | 1 | 1 | 2
Influenza (Infections and infestations) | 0 | 3 | 0 | 2 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 2 | 1 | 0 | 3
Sinusitis (Infections and infestations) | 1 | 0 | 2 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 2
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Clostridial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Vaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 6 | 3 | 4 | 3 | 3
Dizziness (Nervous system disorders) | 1 | 1 | 2 | 1 | 0 | 0
Migraine (Nervous system disorders) | 3 | 0 | 0 | 1 | 0 | 0
Cervical root pain (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Syncope vasovagal (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 5 | 3 | 3 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 2 | 2 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 4 | 0 | 3 | 1 | 3
Fatigue (General disorders) | 1 | 1 | 1 | 2 | 0 | 2
Pain (General disorders) | 1 | 2 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 2 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Infusion site erythema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Infusion site pruritus (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 2
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 3 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
Platelet count increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood pressure decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Occult blood positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 0 | 0 | 0 | 2
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intermittent claudication (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Transmission of drug via semen (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The count of patients with any nonserious adverse events (NAE) excludes patients who only had NAE that occurred in <=5% of patients. This information may vary from existing approved labeling and publications due to the requirement of this website.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the only disclosure restriction on the PI is that the sponsor has 60 days to review results communications prior to public release and can embargo communications regarding trial results for a period that does not exceed 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.